CLINICAL TRIAL: NCT07182435
Title: A Phase 1 Clinical Trial of Personalized mRNA Tumor Vaccine RH125 in Patients With Advanced or Metastatic Solid Tumors Evaluating the Safety, Tolerability, and Efficacy
Brief Title: Exploratory Clinical Study of Personalized mRNA Tumor Vaccine RH125 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RH125-0-01
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- escalation doses between 100μg, 150μg or 200μg of RH125 with or withoout PD-1 blockers (Experimental)
  Interventions: Biological: personalized neoantigen mRNA tumor vaccine

INTERVENTIONS:
Biological: personalized neoantigen mRNA tumor vaccine — RH125 is a personalized neoantigen mRNA tumor vaccine which is constructed based on the results of patients' neoantigen sequencing.

SUMMARY:
This is a Phase 1 clinical study investigating RH125 as monotherapy or in combination therapy in patients with locally advanced or metastatic solid tumors who failed standard treatment, or were intolerant to standard treatment, or declined standard treatment. The aim of the study is to evaluate the tolerability, safety, immunogenicity, and preliminary efficacy of RH125 monotherapy or combination with PD-1 blocker.

DETAILED DESCRIPTION:
This study will be divided into monotherapy dose escalation and combination therapy dose escalation phases. Each phase requires the enrollment of 12-18 subjects, with a total of 24-36 subjects to be enrolled in the entire study. Both the monotherapy dose escalation and combination therapy dose escalation will involve 3 dose levels, which are 100 μg, 150 μg, and 200 μg respectively. A "3+3" design will be adopted, and the Dose-Limiting Toxicity (DLT) observation period will be 21 days for both phases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged from 18 to 70 years old.
2. Patients with histologically and radiologically confirmed locally advanced or metastatic solid tumors that are not suitable for curative surgical treatment, Eligible patients must have experienced disease progression following standard antitumor therapy or be unable or unwilling to receive standard treatments. Patients in the combination therapy group are suitable for PD-1 blockers therapy judged by the investigator .
3. Patients must hava at least one measureble disease per RECIST 1.1.
4. Patients must have a fresh tumor lession sample for sequencing and test of expression of PD-1(22c3,only for patients in the combination therapy group .)
5. ECOG performance status of 0 or 1
6. Life expectancy of at least 6 months.
7. Adequate organ and hematologic function, with no severe dysfunction of the heart, lungs, liver, kidneys, or immune system, based on the following laboratory values:

1). Hematology: ANC ≥ 1.5 × 10⁹/L, PLT ≥ 100 × 10⁹/L, HGB ≥ 100 g/L. Within one week before screening, the subject must not have received blood or platelet transfusions, G-CSF, or erythropoietin (EPO); 2). Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula); 3). Liver function: AST and ALT ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver cancer or liver metastases); TBIL ≤ 1.5 × ULN (patients with Gilbert's syndrome: TBIL < 3 × ULN); 4). Coagulation: INR ≤ 1.5 × ULN or APTT ≤ 1.5 × ULN (except for patients on anticoagulants).

8.. Male subjects with reproductive potential and female subjects of childbearing potential agree to use effective contraception from the time of informed consent until 6 months after the last dose of investigational drug.

Women of childbearing potential include premenopausal women and those within 2 years post-menopause.

A negative serum pregnancy test is required within 7 days before the first dose of the investigational product.

Exclusion Criteria:

1. Having active malignant tumors within 2 years before the first administration, except for any locally curable tumors that have received radical treatment (e.g., resected basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix or breast);
2. Presecne of central nervous system metastases, carcinomatous meningitis, or primary central nervous system tumors.
3. Results of predicted neoantigen epitopes is less than 5.
4. Having received other anti-tumor treatments (such as chemotherapy, endocrine therapy, targeted therapy, immunotherapy, radiotherapy, or tumor embolization) within 4 weeks before the first vaccination; for oral fluoropyrimidines and small-molecule targeted drugs, the interval required is more than 2 weeks or 5 half-lives of the drug, whichever is longer.
5. Clinically significant residual toxicity (≥ grade 2 per CTCAE v5.0) from previous treatment (including systemic therapy, radiotherapy, or surgery), except for alopecia, hyperpigmentation, or other AEs deemed by the investigator not to affect study safety and where recovery to grade ≤1 is not required.
6. Prior one marrow transplantation, allogeneic hematopoietic stem cell transplantation or solid organ transplantation
7. Patients who need to take immunosuppressants regularly within 4 weeks before the first vaccination and during the clinical study, including but not limited to the following situations: those with severe asthma, autoimmune diseases or immunodeficiency, those receiving immunosuppressive drug therapy, or those with a known history of primary immunodeficiency; however, subjects with the following diseases are allowed to undergo further enrollment screening: type I diabetes with good control, hypothyroidism with good control requiring only hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia), or subjects whose condition is not expected to relapse without external triggers.
8. Clinically diagnosed active bacterial or fungal infections; having active tuberculosis or a history of tuberculosis.
9. Active hepatitis B virus (HBV) infection (defined as HBsAg positive and HBV-DNA > ULN), hepatitis C virus (HCV) infection (defined as HCV-Ab positive and HCV-RNA positive), human immunodeficiency virus (HIV) infection (HIV-Ab positive) or treponema pallidum(TP) infection.
10. Severe cardiovascular diseases occurring within 2 years before the first administration, including but not limited to: stable angina pectoris with functional class III-IV; unstable angina pectoris or myocardial infarction; NYHA class III-IV congestive heart failure; severe arrhythmias requiring drug treatment.
11. A history of substance abuse, or clinical, psychological, or social factors that may affect informed consent or the conduct of the study; a history of mental illness.
12. A history of allergies to previous vaccinations, allergies to any component of the investigational product, a history of severe allergies to food or drugs, or other potential allergies to immunotherapy as deemed by the investigator.
13. Pregnant or lactating women.
14. Participation in other interventional clinical studies within 12 weeks before the first vaccination, except for participation in observational (non-interventional) clinical studies or being in the survival follow-up phase of interventional studies.
15. Vaccination of any type within 28 days before administration.
16. Subjects deemed unsuitable for enrollment by the investigator or who may be unable to complete the trial for other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLT) | From Day 1 to Day 21 after the first dose
Number of Participants with Adverse Events per CTCAE 5.0 | Up to approximately 24 months
Immunogenicity of a personalized cancer vaccine as measured by interferon-γ secreting T lymphocytes in peripheral blood mononuclear cells (PBMCs) using ELISpot | Up to approximately 24 months
Serious adverse events as graded by CTCAE v5.0 | Up to approximately 24 months
adverse event of special interest as graded by CTCAE v5.0 | Up to approximately 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the proportion of participants whose best overall response is complete response (CR) or partial response (PR) per RECIST 1.1.
Disease Control Rate(DCR) | Up to approximately 24 months
  ORR is defined as the proportion of participants whose best overall response is complete response (CR) , partial response (PR) or stable disease (SD) per RECIST 1.1.
Rime to response(TTR) | Up to approximately 24 months
  TTR is defined as time to the first tumor response (complete response (CR) or partial response (PR)) per RECIST 1.1.
Duration of Response(DoR) | Up to approximately 24 months
  DoR is defined as time from first tumor response (partial or complete) until either radiological disease progression, clinical/symptomatic disease progression or death (whichever is sooner) per RECIST 1.1.
Progression Free Survival(PFS) | Up to approximately 24 months
  PFS is defined as time between the date of first dose and the date of either radiological disease progression per RECIST 1.1, clinical/symptomatic disease progression or death (whichever is sooner).
Overall Survival(OS) | Up to approximately 24 months
  OS is defined as time between the date of the first dose of study drug and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center; Jianhua Chang, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No